CLINICAL TRIAL: NCT02386605
Title: Motivational Negative Symptoms in Schizophrenia: Intervention and Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1851-W
Record Dates: First submitted 2015-01-23; First posted 2015-03-12 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: recovery; rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Motivational Interviewing Treatment group
  Interventions: Behavioral: Motivational Interviewing and Cognitive Behavioral Therapy
- Control (Active Comparator): Relaxation Skills Training group
  Interventions: Behavioral: Relaxation Skills

INTERVENTIONS:
Behavioral: Motivational Interviewing and Cognitive Behavioral Therapy — group-based recovery-oriented Motivational Interviewing combined with cognitive-behavioral therapy to target the negative symptoms of schizophrenia
  Arms: Treatment
Behavioral: Relaxation Skills — Relaxation and mindfulness skills training group for comparison condition for negative symptoms of schizophrenia
  Arms: Control

SUMMARY:
Negative symptoms significantly interfere with daily functioning among individuals with schizophrenia. They are strongly related to functional impairments [1] and contribute to the poor community outcomes of Veterans with schizophrenia. Motivational negative symptoms interfere with obtaining and maintaining employment [2], forming social relationships[3] and living independently [4]. Developing treatments to effectively reduce negative symptoms is important to achieve improvements in daily functioning. Recent empirical studies report that psychosocial interventions for negative symptoms can have a moderate to large effect size on community functioning and negative symptom severity. However, the treatments that have been utilized so far are either cognitive-behavioral therapy interventions that require over a year of weekly individual sessions and thus are very resource- and time-intensive, or they are skills-training groups that do not address any of the cognitive and motivational aspects of negative symptoms. Although group treatments are increasingly hailed as the gold standard for schizophrenia, there is currently no group intervention explicitly for motivational negative symptoms and functional deficits. Furthermore, treatment development and clinical trials are increasingly reliant on neurophysiological measures of clinical severity and treatment response and so far there are not identified negative symptom biomarkers.

The current CDA proposal will test a group-based treatment based on established motivational enhancement (MI) techniques, augmented with cognitive-behavioral approaches, compared to an active control group treatment, for improving motivational negative symptoms in Veterans with schizophrenia. I will assess the efficacy of MI with measures from two outcome domains: 1) negative symptoms (clinical ratings) and 2) functional outcomes (real-world improvements in social, instrumental, and independent living). I will assess the relationship between these outcomes and neurophysiological biomarkers (pupillometry and electroencephalography (EEG)). Participants will be randomly assigned to the MI treatment or a control treatment for weekly 1-hour sessions for 12 weeks. The assessment battery will be administered at baseline, at completion of treatment, and at 6-month follow-up. The investigators will enroll 60 Veterans with schizophrenia that are low functioning and have high negative symptoms across the 4 years of the study.

This proposal is designed to examine group-based MI for reducing negative symptoms and improving functioning in key domains (i.e., interpersonal, instrumental, and independent living skills). Moreover, it will thoroughly investigate biomarkers of negative symptoms with pupillometry and EEG. The development and evaluation of this recovery- oriented group MI treatment for Veterans with disabling negative symptoms will yield results that can inform larger treatment trials and neurophysiological measurement of negative symptoms in Veterans with schizophrenia.

DETAILED DESCRIPTION:
Despite significant advances in pharmacological treatments for schizophrenia (SCZ), the rate of disability among Veterans diagnosed with SCZ remains high. Functional disability among Veterans with SCZ creates a huge and costly burden on the national VA healthcare system, and interferes with community integration and quality of life. In particular, SCZ is associated with low rates of employment, few social relationships, and poor independent living skills. The negative symptoms of SCZ (i.e. avolition, anhedonia, asociality) are primary determinants of functional impairments, and they have no validated treatments. Extensive work has been devoted to treating positive symptoms and cognitive deficits, but much less has been done to develop pharmacological and psychosocial treatments for negative symptoms. Developing such interventions is a critical public health goal, as it would benefit one of the largest groups of disabled Veterans.

The recently-emerging recovery-oriented approach to serious mental illness reflects a fundamental shift from a focus on symptom reduction to a focus on patients' goals and community functioning. Developing treatments for negative symptoms to augment community functioning is a strong reflection of this shift. Importantly, preliminary research suggests that motivational negative symptoms respond to novel evidence-based psychosocial interventions. The primary goal of this proposal is to adapt and implement a recovery-oriented evidence-based intervention, Motivational Interviewing (MI), for the treatment of motivational negative symptoms in Veterans with SCZ. MI, originally developed for substance use disorders, is effective to increase commitment to new behaviors in a range of areas including treatment adherence, exercise, gambling, and depression. Importantly, it has been shown to be applicable to Veterans with psychosis, but it is not known if MI can reduce functional deficits that are attributable to motivational negative symptoms.

More specifically, the scientific goals of this proposal are to: 1) evaluate the efficacy of a group-based MI intervention on motivational negative symptoms for Veterans with SCZ, and 2) to examine potential biomarkers of negative symptoms and treatment response. I will assess the efficacy of MI with measures from two outcome domains: 1) negative symptoms (clinical ratings) and 2) functional outcomes (real-world improvements in social, instrumental, and independent living). I will assess the relationship between these outcomes and neurophysiological biomarkers (pupillometry and electroencephalography (EEG)). To address these questions, 60 Veterans with SCZ who have at least moderate levels of motivational negative symptoms will be randomly assigned in a 1:1 ratio to MI or a standard treatment (relaxation skills training). Both treatments will consist of weekly 60-min group sessions for twelve weeks. The assessment will be administered at baseline, at completion of treatment, and at 6-month follow-up.

Specific Aim #1: To adapt the existing MI approach for group-based MI treatment for Veterans with SCZ.

Specific Aim #2: To examine the treatment effects of MI compared to the control procedure on motivational negative symptoms and functional outcomes.

Hypothesis 2a: Individuals who receive MI will have significant improvements in motivational negative symptoms, compared to those who receive the control.

Hypothesis 2b: Individuals who receive MI will have significant improvements in aspects of functioning including social, instrumental, and independent living domains, compared to those who receive the control.

Specific Aim #3: To examine neurophysiological biomarkers (i.e., EEG and pupillometry) of motivational negative symptom severity and treatment response.

Hypothesis 3a: At baseline, subjects with more negative symptoms at baseline will have more aberrant EEG and pupillary measures.

Hypothesis 3b: For subjects in the treatment group, change in the biomarkers (toward normalization) over study duration will correlate with treatment related improvement in motivational negative symptoms.

Exploratory Aim: To explore a causal model by examining whether MI improves defeatist beliefs compared to a control procedure.

Although MI is a well-established intervention for a range of clinical populations and conditions, the proposed project will be the first examination of MI in a group format for motivational negative symptoms in SCZ. If validated, it could be disseminated throughout the VA for other patient populations with motivational and functional deficits (e.g., traumatic brain injury, post-traumatic stress disorder). Therefore, this CDA application will facilitate my research independence and provide me with a unique combination of skills that will equip me to be a local professional resource and long-term VA researcher.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* No medication changes in the past six weeks
* No psychiatric hospitalization in the past three months
* No changes in housing in the past two months

Exclusion Criteria:

* Neurological disorder
* seizures
* history of serious head injury
* substance dependence in the past 6 months or abuse in the past month
* being insufficiently fluent in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena F Reddy, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy LF, Glynn SM, McGovern JE, Sugar CA, Reavis EA, Green MF. A Novel Psychosocial Intervention for Motivational Negative Symptoms in Schizophrenia: Combined Motivational Interviewing and CBT. Am J Psychiatry. 2023 May 1;180(5):367-376. doi: 10.1176/appi.ajp.20220243. Epub 2023 Mar 9. PMID 36891649

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 99 enrolled participants 79 met inclusion criteria and were randomized to one of the two conditions
Period: Overall Study
Arm/Group | Treatment | Control
Started | 41 | 38
Completed | 34 | 28
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 41 | 38 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 38 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (8.8) | 54.1 (8.2) | 54.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 39 | 36 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 20 | 43
  White | 13 | 14 | 27
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 38 | 79

OUTCOME MEASURES:

1. Primary Outcome: Strauss-Carpenter Level of Function Scale
Description: This scale is a 43-item report of a patient's behavior and functioning across the following domains: physical functioning (e.g., vision, hearing), personal care skills (e.g., eating, grooming), interpersonal skills (e.g., initiating, accepting, and maintaining social contacts; effectively communicating), social acceptability (e.g., absence of verbal and physical abuse, absence of repetitive behaviors), community activities (e.g., shopping, using the telephone, paying bills, use of leisure time, use of public transportation), and work skills (e.g., employable skills, level of supervision, punctuality). Each item is rated on a 5 point likert scale. A functional skill composite is created by summing the interpersonal relationships, activities, and work skills domains. The range for the summary score was 64 - 120, with higher scores indicating better functioning.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 41 | 38
score on a scale | 97.69 (13.8) | 94.56 (11.5)

2. Primary Outcome: Clinical Assessment Interview for Negative Symptoms
Description: The CAINS is a 13-item instrument that yields two subscales which measure the two primary negative symptom factors: Motivation and Pleasure (MAP) which measures experiential negative symptoms and Expression which measures the expressive negative symptoms. The MAP was used as a primary dependent variable, it includes 9 items rated 0-4 and yields a mean subscale (0-4). Higher scores reflect greater impairment.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 41 | 38
score on a scale | 2.1 (.82) | 1.3 (.78)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02386605/Prot_SAP_000.pdf